CLINICAL TRIAL: NCT00207597
Title: A Clinical Trial of Primary Prophylaxis Against Joint Disease in Children With Severe Hemophilia
Brief Title: Joint Outcome Study
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Other Study IDs: CDC-NCBDDD-1455; U27/CCU812106
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

SUMMARY:
This study examines the progression of joint disease in children with hemophilia assigned to either standard treatment or enhanced therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hemophilia A
* factor level less than 2%

Exclusion Criteria:

* More than 2 bleeds into the same joint

Ages: 1 Year to 30 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64
Dates: Start 1995-09; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn J Manco-Johnson, MD, Principal Investigator — University of Colorado, Denver

REFERENCES:
- [Derived] Warren BB, Jacobson L, Kempton C, Buchanan GR, Recht M, Brown D, Leissinger C, Shapiro AD, Abshire TC, Manco-Johnson MJ; Joint Outcome Study Group Investigators. Factor VIII prophylaxis effects outweigh other hemostasis contributors in predicting severe haemophilia A joint outcomes. Haemophilia. 2019 Sep;25(5):867-875. doi: 10.1111/hae.13778. Epub 2019 May 21. PMID 31115111
- [Derived] Manco-Johnson MJ, Abshire TC, Shapiro AD, Riske B, Hacker MR, Kilcoyne R, Ingram JD, Manco-Johnson ML, Funk S, Jacobson L, Valentino LA, Hoots WK, Buchanan GR, DiMichele D, Recht M, Brown D, Leissinger C, Bleak S, Cohen A, Mathew P, Matsunaga A, Medeiros D, Nugent D, Thomas GA, Thompson AA, McRedmond K, Soucie JM, Austin H, Evatt BL. Prophylaxis versus episodic treatment to prevent joint disease in boys with severe hemophilia. N Engl J Med. 2007 Aug 9;357(6):535-44. doi: 10.1056/NEJMoa067659. PMID 17687129